CLINICAL TRIAL: NCT00028925
Title: Phase II Trial of Oral Topotecan and Intravenous Carboplatin With G-CSF (Filgrastim) Support in Previously Untreated Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Combination Chemotherapy With or Without Filgrastim in Treating Patients With Previously Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0027; NCI-2012-02441 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000069147 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-06-30 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Experimental): Patients receive oral topotecan once daily on days 1-5, carboplatin IV over 30 minutes on day 5, and filgrastim (G-CSF) subcutaneously once daily beginning on day 6 or 7 and continuing for up to 10 days or until blood counts recover.
  Treatment for all patients repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression limited to CNS only interrupt chemotherapy to have whole-brain radiotherapy (WBRT). Once WBRT is complete, chemotherapy resumes.
  Quality of life is assessed at baseline and at the beginning of each course of chemotherapy.
  Patients are followed every 3 months for 2 years and then every 6 months for 3 years.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: topotecan hydrochloride; Radiation: WBRT
- Regimen B (Experimental): Patients receive topotecan and carboplatin as in regimen A. Patients are evaluated after the first 3-week course of chemotherapy. If no patient experiences unacceptable toxicity or febrile neutropenia, the next 33 patients receive treatment as in regimen B; otherwise, patients receive treatment as in regimen A.
  Treatment for all patients repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression limited to CNS only interrupt chemotherapy to have whole-brain radiotherapy (WBRT). Once WBRT is complete, chemotherapy resumes.
  Quality of life is assessed at baseline and at the beginning of each course of chemotherapy.
  Patients are followed every 3 months for 2 years and then every 6 months for 3 years.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: topotecan hydrochloride; Radiation: WBRT

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: topotecan hydrochloride
Radiation: WBRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to compare the effectiveness of combination chemotherapy with or without filgrastim in treating patients who have extensive-stage small cell lung cancer that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerability of topotecan and carboplatin with or without filgrastim (G-CSF) in patients with extensive stage small cell lung cancer.
* Determine response and survival rates in patients treated with these regimens.

OUTLINE: This is a multicenter study. The first 12 patients are assigned to 1 of 2 treatment regimens (6 per regimen). The next 33 patients receive treatment based on the toxicity experienced by the first 12.

Regimen A:

* Patients receive oral topotecan once daily on days 1-5, carboplatin IV over 30 minutes on day 5, and filgrastim (G-CSF) subcutaneously once daily beginning on day 6 or 7 and continuing for up to 10 days or until blood counts recover.
* Patients are evaluated after the first 3-week course of chemotherapy. If no patient experiences unacceptable toxicity or febrile neutropenia, or no more than 1 patient experiences an absolute neutrophil count of less than 500/mm3 for more than 5 days, the next 6 patients begin treatment on regimen B. Otherwise, all patients receive treatment as in regimen A.

Regimen B:

* Patients receive topotecan and carboplatin as in regimen A.
* Patients are evaluated after the first 3-week course of chemotherapy. If no patient experiences unacceptable toxicity or febrile neutropenia, the next 33 patients receive treatment as in regimen B; otherwise, patients receive treatment as in regimen A.

Treatment for all patients repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression limited to CNS only interrupt chemotherapy to have whole-brain radiotherapy (WBRT). Once WBRT is complete, chemotherapy resumes.

Quality of life is assessed at baseline and at the beginning of each course of chemotherapy.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 49 patients will be accrued for this study within 13.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung cancer

  * Previously untreated with chemotherapy
  * No mixed histology
* Metastatic disease outside the chest

  * Contralateral supraclavicular or hilar nodes that cannot be included in a single radiation port OR
  * Cytologically proven malignant pleural effusion
* Measurable disease
* No untreated CNS metastases

  * CNS metastases treated with whole-brain radiotherapy (WBRT) allowed after completion of WBRT

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* AST no greater than 5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* Bilirubin no greater than 1.5 times ULN OR
* Direct bilirubin no greater than ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No uncontrolled angina pectoris
* No congestive heart failure within the past 3 months unless ejection fraction is greater than 40%
* No uncontrolled cardiac arrhythmias
* No myocardial infarction within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant infection
* No hypersensitivity to E. coli-derived proteins
* No other malignancy within the past 3 years except non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 5 years since prior chemotherapy for another malignancy
* No prior nitrosoureas

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior thoracic radiotherapy
* At least 1 day since prior palliative radiotherapy (except to chest)
* No more than 3 fractions to chest for superior vena cava syndrome allowed
* No concurrent radiotherapy (including thoracic radiotherapy)

Surgery:

* More than 3 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-11; Primary Completion 2005-11 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James R. Jett, MD, Study Chair — Mayo Clinic
Locations (24):
- United States (23):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Wichita Community Clinical Oncology Program, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Bryce AH, Mattar B, Hillman SL, Adjei AA, Kugler JW, Rowland K Jr, Wender DB, Soori G, Perez EA, Jett JR. Phase II trial of oral topotecan and intravenous carboplatin with G-CSF support in previously untreated patients with extensive stage small cell lung cancer: A North Central Cancer Treatment Group Study. Am J Clin Oncol. 2010 Aug;33(4):353-7. doi: 10.1097/COC.0b013e3181b0c27f. PMID 19935387